CLINICAL TRIAL: NCT05522881
Title: The Registry Study of Genetic Alterations of Oropharyngeal Cancer in Taiwan
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T1322
Record Dates: First submitted 2022-08-23; First posted 2022-08-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
Keywords: human papillomavirus; oropharyngeal squamous cell carcinoma; next-generation sequencing; precision medicine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — One H&E-stained slide, and at least 10 unstained tissue on non-coated slides (5 um thickness) for cancer panel-based NGS analysis.20 unstained tissue on non-coated slides (4 um thickness) will be required for HPV genotyping testing.
  20 ml Cell-Free DNA blood will be collected from the subjects within two weeks of the study registration. Of the treatment-naïve group, 20 ml blood specimens will be additionally collected at week 4 and 8 after the curative therapy is completed then every 6 months until the study withdrawal or tumor recurrence. For all subjects receiving the curative therapy, 20 ml of blood specimen will be collected when tumor recurrence is diagnosed at follow-up after the study registration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- HPV positive-Post treatment: The subject has received any anti-cancer treatment with pathological report of squamous cell carcinoma of oropharynx (soft palate, tonsil, base of tongue, pharyngeal wall, uvula or vallecula) and positive p16 immunohistochemical staining.
- HPV negative-Post treatment: The subject has received any anti-cancer treatment with pathological report of squamous cell carcinoma of oropharynx (soft palate, tonsil, base of tongue, pharyngeal wall, uvula or vallecula) and negative p16 immunohistochemical staining.
- HPV positive-Treatment-naïve: The subject has received no anti-cancer treatment with pathological report of squamous cell carcinoma of oropharynx (soft palate, tonsil, base of tongue, pharyngeal wall, uvula or vallecula) and positive p16 immunohistochemical staining.
- HPV negative-Treatment-naïve: The subject has received no anti-cancer treatment with pathological report of squamous cell carcinoma of oropharynx (soft palate, tonsil, base of tongue, pharyngeal wall, uvula or vallecula) and negative p16 immunohistochemical staining.
- reference subgroup: 60 patients with head and neck SCC (excluding OPSCC)
- recurrence subgroup: pairs of primary and recurrent tumors (at the first distal or local recurrence) of head and neck SCC

SUMMARY:
We will use the next-generation sequencing (NGS) technology to identify genomic alterations of Taiwanese HPV positive and negative oropharyngeal squamous cell carcinoma (OPSCC) for novel biomarker development and the study design of potential clinical trials or translational research.

DETAILED DESCRIPTION:
In the past decade, next-generation sequencing (NGS) technology has enabled cancer genome sequencing in screening and searching for new cancer genes in an efficient manner. This massive sequencing technique not only help to identify new altered genes for novel biomarker development, but also reveal gene alterations sensitive or resistant to specific therapies. Because the difference of genomic profiling between Taiwanese HPV positive and negative OPSCC is not clear yet, we propose this multi-center research project to address this issue. In this study, we will collect tumor tissues and clinical information from patients with OPSCC and create a platform for data storage and sharing.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20 and above
2. Pathological reported as squamous cell carcinoma of head and neck
3. Available p16 immunohistochemical staining status (restricted to the OPSCC subgroup)
4. Participants have both archival tumor tissues from the primary head and neck SCC and from the first recurrent tumor (for the recurrence subgroup)
5. Recurrence status is defined as the reappearance of the disease occurring more than 6 months following curative surgery and/or chemoradiotherapy in the recurrence subgroup
6. Willingness to provide archival or newly obtained tumor tissues for current study proposal
7. Life expectancy more than 3 months
8. Patients fully understand the protocol with the willingness to have regular follow-up

Exclusion criteria

1. Inability to cooperate by providing a complete medical history
2. No available tumor tissues for genetic testing
3. Undesirable compliance
4. Having a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To enroll a total of 410 patients with head and neck SCC
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To enroll a total of 300 patients with OPSCC who fit the criteria of this study in the enrolled period | 5 years of proposed observation period
  To enroll a total of 300 patients with OPSCC who fit the criteria of this study in the enrolled period

SECONDARY OUTCOMES:
To perform next generation sequencing analysis of OPSCC tumor tissues | 5 years of proposed observation period
  To perform next generation sequencing analysis of OPSCC tumor tissues
Collect clinical data of OPSCC | 5 years of proposed observation period
  To correlate with the clinical characteristics and treatment outcomes of patients with the genetic profile in Taiwan.
To compare the difference of the genetic and molecular profiles among patients with HPV positive and negative OPSCC | 5 years of proposed observation period
  To compare the difference of the genetic and molecular profiles among patients with HPV positive and negative OPSCC
To compare the difference of genetic and molecular profiles between early (stage I and II) and advanced stage (stage III and IV) of HPV positive OPSCC | 5 years of proposed observation period
  To compare the difference of genetic and molecular profiles between early (stage I and II) and advanced stage (stage III and IV) of HPV positive OPSCC

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, MD, PhD, Principal Investigator — National Taiwan University Hospital; Shang-Hung Chen, MD, PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (7):
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Pei-Jen Alex Lou, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided